CLINICAL TRIAL: NCT03188770
Title: PRactice of VENTilation in Critically Ill Patients in Middle-Income Countries (PRoVENT-iMIC) - an International Multicenter Service Review Focusing on ICUs in Asia
Brief Title: Practice of Ventilation in Middle-Income Countries
Acronym: PRoVENT-iMIC
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PRoVENT-iMIC
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Mechanical Ventilation; Respiratory Distress Syndrome, Adult; Acute Respiratory Failure
Keywords: Middle-income countries
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical Ventilation: Patients under mechanical ventilation in the ICU

SUMMARY:
The purpose of this international, multicenter service review is to describe and compare ventilation management in patients at risk of acute respiratory distress syndrome (ARDS) versus patients not at risk and patients with established ARDS, and to ascertain whether certain ventilator settings and ventilation parameters are associated with pulmonary complications or development of ARDS after start of ventilation in patients in intensive care units (ICUs) in Asian countries.

Participating centers will include adult patients undergoing mechanical ventilation in the ICU during a 28-day period. Patients' data will be collected during the first 7 days in the ICU, or until ICU discharge. Follow up is until ICU discharge. The primary outcome includes two main ventilator settings, i.e., tidal volume and the level of positive end-expiratory pressure. Secondary endpoints are development of ARDS in patients without ARDS at the onset of mechanical ventilation, worsening of ARDS in patients with ARDS at the onset of mechanical ventilation, pulmonary infection, other pulmonary complications, need for tracheostomy, duration of ventilation, length of ICU stay and ICU mortality.

DETAILED DESCRIPTION:
Rationale: scarce information exists on management of mechanical ventilation in intensive care unit (ICU) patients in low- and middle-income countries.

Objective:The primary objective is to describe and compare ventilation management in patients at risk of ARDS versus individuals not at risk, and patients with established ARDS, and to ascertain whether certain ventilation settings are associated with a higher incidence of developing ARDS in patients in ICUs in Asia. PRoVENT-iMIC secondary objectives are to determine the epidemiological characteristics and clinical outcomes of patients at risk of ARDS in ICUs in Asia according to the ventilation practice applied.

Primary hypothesis: a large proportion of patients at risk of ARDS in ICUs in Asia do not receive so-called protective ventilation, defined as tidal volume < 8 ml/kg predicted body weight and a level of positive end-expiratory pressure of at least 5 cm H2O.

Secondary hypothesis: in ICUs in Asia a large proportion of patients is at risk of ARDS, as stratified by a Lung Injury Prediction Score of ≥4.

Study design: an international multicenter service review focusing on ICUs in selected middle-income Asian countries.

Population: consecutive intubated and ventilated ICU patients.

Methods: Patients in participating ICUs will be screened daily during a 28-day period. A registry of limited demographic data will be compiled on all screened patients. Collection of ventilation characteristics is restricted to the first three days. The first seven days or up to death, whichever comes first, will be used for collection of patient demographics (on day of admission), development of ARDS and other pulmonary complications. All patients will be followed until ICU-discharge to determine length of stay in ICU and ICU mortality. The inclusion period will be flexible for participating centers and determined at a later stage together with the study-coordinator. Data will be coded by a patient identification number of which the code will be kept safe at the local sites. The data will be transcribed by local investigators onto an internet based electronic case report form (https://www.project-redcap.org).

Centers: about 60 Asian ICUs from ten countries are expected to participate in this international multicenter study. Each participating center will recruit ~ 50 patients.

Ethics Approval: The Oxford Tropical Research Ethical Committee has evaluated the study and considered it exempt from ethical review on the 1st of June 2017. National coordinators will be responsible for clarifying the need for ethics approval and applying for this where appropriate according to local policy. Centers will not be permitted to record data unless ethics approval or an equivalent waiver is in place.

Monitoring: Due to the observational nature of the study, a Data Safety and Monitoring Board is not necessary.

Sample Size Calculation: a formal sample size calculation was not performed, seen the largely descriptive character of this investigation. 3000 patients are expected to be enrolled in the study period, which will be sufficient to test the hypotheses.

Statistical Analysis: Patient characteristics will be compared and described by appropriate statistics. Student's t-test or Mann-Whitney U-tests are used to compare continuous variables and chi-squared tests are used for categorical variables. Data are expressed as means (SD), medians (interquartile range) and proportions as appropriate. Comparisons between and within groups are performed using one-way ANOVA and post-hoc analyses for continuous variables.

The primary analysis concerns the determination of (variation of) tidal volume and PEEP levels in patients without ARDS. These are compared between predefined patient groups: patients at no risk for ARDS, patients at risk for ARDS, patients with mild ARDS, and patients with moderate or severe ARDS.

To identify potential factors associated with outcome like development of ARDS, or worsening of ARDS, development of pulmonary complications, duration of ventilation, or death, univariate analyses are performed. A multivariate logistic regression model is used to identify independent risk factors. A stepwise approach is used to enter new terms into the model, with a limit of p < 0.2 to enter the terms. Time to event variables are analyzed using Cox regression and visualized by Kaplan-Meier.

Organization: The study is conducted by the PROtective VEntilation Network (PROVENet). National co-ordinators will lead the project within individual nations and identify participating hospitals, translate study paperwork, distribute study paperwork and ensure necessary regulatory approvals are in place. They provide assistance to the participating clinical sites in trial management, record keeping and data management. Local coordinators in each site will supervise data collection and ensure adherence to Good Clinical Practice during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an ICU participating in this study
* Intubated in the ICU, or in the emergency room, general ward, or operation room before the present ICU admission

Exclusion Criteria:

* Age < 18 years
* Patients under invasive mechanical ventilation previous to the 28-day period of inclusion
* Patients transferred from another hospital under invasive mechanical ventilation
* Receiving only non-invasive ventilation (i.e., patient never received invasive ventilation during the present admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive intubated and ventilated intensive care unit patients
Sampling Method: Probability Sample
Enrollment: 1315 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Tidal volume size | Day 1 to Day 3 from initiation of mechanical ventilation
  Tidal volume size in milliliters per kilogram of predicted body weight
Positive end-expiratory pressure | Day 1 to Day 3 from initiation of mechanical ventilation
  Pressure in cm of water

SECONDARY OUTCOMES:
Patients at risk of ARDS | On the date of inclusion
  Risk of ARDS is stratified using the Lung Injury Prediction Score.
Inspired Oxygen Concentration | Day 1 to Day 3 from initiation of mechanical ventilation
  expressed as fraction of inspired oxygen
Plateau pressure | Day 1 to Day 3 from initiation of mechanical ventilation
  Pressure in cm of water
Peak pressure | Day 1 to Day 3 from initiation of mechanical ventilation
  Peak away pressure in cm of water
Driving pressure | Day 1 to Day 3 from initiation of mechanical ventilation
  pressure in cm of water
Respiratory Rate | Day 1 to Day 3 from initiation of mechanical ventilation
  in breaths per minute
Minute Volume | Day 1 to Day 3 from initiation of mechanical ventilation
  expressed as liters per minute
Development of ARDS | From date of inclusion until the date of first documented development of ARDS or date of ICU discharge or death from any cause, whichever came first, assessed up to 7 days
  Development of ARDS in patients without ARDS at the onset of mechanical ventilation. Patients are defined as having ARDS if they meet the Berlin criteria for ARDS
Worsening of ARDS | From date of inclusion until the date of first documented worsening of ARDS or date of ICU discharge or death from any cause, whichever came first, assessed up to 7 days
  Defined as any worsening in the degree of severity according to Berlin criteria.
Pulmonary infection | From date of inclusion until the date of first documented pulmonary complication or date of ICU discharge or death from any cause, whichever came first, assessed up to 7 days
  defined as need of new antibiotics in the presence of new or changed lung opacities on chest X-ray and/or new or changed sputum plus at least one of the following criteria: 1) temperature > 38.3 ºC; or 2) WBC count > 12,000
Other Pulmonary complications | From date of inclusion until the date of first documented pulmonary complication or date of ICU discharge or death from any cause, whichever came first, assessed up to 7 days
  pneumothorax, pleural effusions, cardiogenic pulmonary edema, new pulmonary infiltrates, and atelectasis
Need for tracheostomy | From date of inclusion until the date of first documented tracheostomy procedure or date of ICU discharge or death from any cause, whichever came first, assessed up to 7 days
  Need for tracheostomy during ICU stay
Length of stay in ICU | Until day 35 from study initiation
  Time between admission and discharge or death
All-cause ICU mortality | Until day 35 from study initiation
  Any death during ICU stay
Duration of mechanical ventilation | Until day 35 from study initiation
  time between orotracheal intubation and successful extubation;note: in case of intermittent MV via a tracheostomy, every day a patient needs MV counts as one extra day of MV, irrespective of duration of MV that specific day; in case of non-invasive ventilation (CPAP and/or BIPAP), the duration will be assessed separated from the assessment of invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Arjen M Dondorp, MD, PhD, Principal Investigator — Mahidol Oxford Research Unit, University of Oxford; Luigi Pisani, MD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Ary Serpa Neto, MD, MSc, Study Chair — Hospital Israelita Albert Einstein
Locations (51):
- Bangladesh (6):
  - Chittagong Medical College Hospital, Chittagong
  - Bangabandhu Sheikh Mujib Medical University, Dhaka
  - BIRDEM General Hospital, Dhaka
  - Dhaka Medical College Hospital, Dhaka
  - Rajshahi Medical College Hospital, Rajshahi
  - Sylhet MAG Osmani Medical College Hospital, Sylhet
- India (3):
  - Ispat General Hospital, Raurkela, Odisha
  - St. John's Medical College, Bangalore
  - Bharati Vidyapeeth Medical College, Pune
- Iran (3):
  - Modarres Hospital, Tehran
  - Pars Hospital, Tehran
  - Masih Daneshvari Hospital, Tehrān
- Malaysia (4):
  - Monash University, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Mohamad Irfan Bin Othman Jailani, Kuala Lumpur
  - International Islamic University Medical Center, Kuantan
- Indira Gandhi Memorial Hospital, Malè, Maldives
- Patan Academy of Health Sciences, Kathmandu, Nepal
- Pakistan (10):
  - Allied Hospital, Faisalābad
  - PIMS, Islamabad
  - Shifa International Hospital, Islamabad
  - Aga Khan University Hospital MICU, Karachi
  - Aga Khan University SICU, Karachi
  - Patel Hospital, Karachi
  - Doctor's Hospital, Lahore
  - National Hospital and Medical Center, Lahore
  - Peoples Medical College Hospital, Nawabshah
  - North West General Hospital, Peshawar
- Sri Lanka (11):
  - Batticaloa Base Hospital, Batticaloa
  - Colombo South Teaching Hospital MICU, Colombo
  - Colombo South Teaching Hospital SICU, Colombo
  - Lanka Hospital, Colombo
  - National Hospital Sri Lanka MICU, Colombo
  - National Hospital Sri Lanka SICU, Colombo
  - Sri Jayawardenepura CTICU, Colombo
  - Sri Jayewardenepura General Hospital GICU, Colombo
  - Karapitiya Teaching Hospital, Galle
  - Jaffna Teaching Hospital, Jaffna
  - Puttlam Hospital, Puttalam
- Thailand (10):
  - Chulalongkorn University Hospital, Bangkok
  - Hospital for Tropical Diseases, Mahidol University, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Sriraj Hospital, Bangkok
  - Vajira Hospital, Bangkok
  - Chiang Mai Hospital Surgical ICU, Chiang Mai
  - Chiang Mai Medical ICU, Chiang Mai
  - Nakornping Hospital, Chiang Mai
  - Prince of Songkla University, Hat Yai
  - Srinakharinwirot University, Ongkharak
- Vietnam (2):
  - National Hospital for Tropical Diseases, Hanoi
  - Oxford University Clinical Research Unit, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Result] Neto AS, Barbas CSV, Simonis FD, Artigas-Raventos A, Canet J, Determann RM, Anstey J, Hedenstierna G, Hemmes SNT, Hermans G, Hiesmayr M, Hollmann MW, Jaber S, Martin-Loeches I, Mills GH, Pearse RM, Putensen C, Schmid W, Severgnini P, Smith R, Treschan TA, Tschernko EM, Melo MFV, Wrigge H, de Abreu MG, Pelosi P, Schultz MJ; PRoVENT; PROVE Network investigators. Epidemiological characteristics, practice of ventilation, and clinical outcome in patients at risk of acute respiratory distress syndrome in intensive care units from 16 countries (PRoVENT): an international, multicentre, prospective study. Lancet Respir Med. 2016 Nov;4(11):882-893. doi: 10.1016/S2213-2600(16)30305-8. Epub 2016 Oct 4. PMID 27717861
- [Derived] Serafini SC, Cinotti R, Asehnoune K, Battaglini D, Robba C, Neto AS, Pisani L, Mazzinari G, Tschernko EM, Schultz MJ; PRoVENT, the PRoVENT-iMiC and ENIO, investigators. Potentially modifiable ventilation factors associated with outcome in neurocritical care vs. non-neurocritical care patients: Rational and protocol for a patient-level analysis of PRoVENT, PRoVENT-iMiC and ENIO (PRIME). Rev Esp Anestesiol Reanim (Engl Ed). 2025 May;72(5):501690. doi: 10.1016/j.redare.2025.501690. Epub 2025 Feb 15. PMID 39961531
- [Derived] Serafini SC, van Meenen DMP, Pisani L, Neto AS, Ball L, de Abreu MG, Algera AG, Azevedo L, Bellani G, Dondorp AM, Fan E, Laffey JG, Pham T, Tschernko EM, Schultz MJ, van der Woude MCE; ERICC; LUNG SAFE; PRoVENT; PRoVENT-iMiC-investigators. Different ventilation intensities among various categories of patients ventilated for reasons other than ARDS--A pooled analysis of 4 observational studies. J Crit Care. 2024 Jun;81:154531. doi: 10.1016/j.jcrc.2024.154531. Epub 2024 Feb 10. PMID 38341938
- [Derived] Pisani L, Algera AG, Serpa Neto A, Ahsan A, Beane A, Chittawatanarat K, Faiz A, Haniffa R, Hashemian R, Hashmi M, Imad HA, Indraratna K, Iyer S, Kayastha G, Krishna B, Moosa H, Nadjm B, Pattnaik R, Sampath S, Thwaites L, Tun NN, Yunos NM, Grasso S, Paulus F, de Abreu MG, Pelosi P, Dondorp AM, Schultz MJ; PRoVENT-iMIC investigators, MORU and the PROVE network. PRactice of VENTilation in Middle-Income Countries (PRoVENT-iMIC): rationale and protocol for a prospective international multicentre observational study in intensive care units in Asia. BMJ Open. 2018 Apr 28;8(4):e020841. doi: 10.1136/bmjopen-2017-020841. PMID 29705765
- See also: Study website — https://sites.google.com/site/proventimic/
- See also: Protective Ventilation Network website — https://sites.google.com/site/proveneteu/

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT03188770/SAP_000.pdf